CLINICAL TRIAL: NCT00414011
Title: Comparison of the Effect of 4th Generation Fluoroquinolones, Gatifloxacin and Moxifloxacin, on Epithelial Healing Following Photorefractive Keratectomy (PRK), A Substudy of: Initial Evaluation of Excimer Laser Keratorefractive Surgery in U.S. Army Personnel (WU # 2335-99)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRAMC WU # 04-2335-99e
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-06

CONDITIONS: Epithelium, Corneal
Keywords: Removal of corneal epithelium followed by excimer laser treatment during prk
MeSH Terms: interventions — Moxifloxacin; Gatifloxacin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin eye drops; 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
  Interventions: Drug: Moxifloxacin
- Gatifloxacin (Experimental): Gatifloxacin eyedrops; 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
  Interventions: Drug: Gatifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
  Arms: Moxifloxacin
Drug: Gatifloxacin — 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
  Arms: Gatifloxacin

SUMMARY:
The purpose of this study is a prospective,double-blinded, randomized trial to compare the rate of healing following PRK after the use of two commercially available 4th generation fluoroquinolones, moxifloxacin and gatifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Manifest refraction spherical equivalent (MSE) of up to -6.00 diopters (D) at the spectacle plane with refractive cylinder up to 3.00D.

Exclusion Criteria:

* Concurrent topical or systemic medications that may impair healing including corticosteroids, antimetabolites, isotretinoin, amiodarone hydrochloride and/ or sumatripin.
* Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Anterior basement membrane dystrophy.
* History of recurrent epithelial erosion.
* Significant dry eye (symptomatic sith Schirmer <5mm at 5 minutes)
* Other corneal epithelial disorder or healing abnormality

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S. BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxifloxacin/Gatifloxacin Treatment: Both eyes were treated. Each participant was randomly assigned to either:
  Group A: Moxifloxacin eyedrops on right eye; Gatifloxacin eyedrops on left eye
  Group B: Gatifloxacin eyedrops on right eye; Moxifloxacin eyedrops on left eye
  Eyedrops were given as 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
Period: Overall Study
Arm/Group | Moxifloxacin/Gatifloxacin Treatment
Started | 40
Completed | 35
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 35 out of 40 participants had complete data for analysis.
Arm/Group | Moxifloxacin/Gatifloxacin Treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.7 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Corneal Epithelial Healing Time
Description: patients' eyes will be observed daily after surgery until the corneal epithelium has completely healed (usually 3 to 4 days)
Time Frame: 3 to 4 days after surgery
Measure: Median (Full Range); unit: days to complete epithelial healing
Units Other Than Participants: eyes
Groups:
- Moxifloxacin: Moxifloxacin eyedrops; 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
- Gatifloxacin: Gatifloxacin eye drops; 1 drop 4 times daily for 1 week or until complete re-epithelization (usually 3-4 days) after surgery
Arm/Group | Moxifloxacin | Gatifloxacin
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
days to complete epithelial healing | 4 (1) [3 to 7] | 4 (1.4) [3 to 9]

ADVERSE EVENTS:
Groups:
- Adverse Events Not Collected: Adverse Events Not Collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All materials that reflects the WRAMC affiliation must be approved and properly cleared before the material is submitted for public dissemination and publication. All publications whereby WRAMC is cited in the bylines will state on the cover page the following sample disclaimer: "The views expressed in this [article, book chapter, speech, presentation, etc.] are those of the author(s) and do not reflect the official policy of the Department of Army, Department of Defense, or U.S. Government."